CLINICAL TRIAL: NCT01528605
Title: The Effects of Lutein and Zeaxanthin Supplementations on Early Age-related Macular Degeneration
Brief Title: Effects of Lutein and Zeaxanthin Supplementation on Early Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaoming Lin, Study Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NNSFC-30872113
Record Dates: First submitted 2011-12-28; First posted 2012-02-08 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Age-related Macular Degeneration
Keywords: lutein; zeaxanthin; age-related macular degeneration; supplementation; macular pigment optical density; visual function; serum concentration
MeSH Terms: conditions — Macular Degeneration | interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): starch in hard shell gelatine capsules
  Interventions: Dietary Supplement: placebo
- Low lutein (Experimental): low lutein group
  Interventions: Dietary Supplement: low lutein
- High lutein (Experimental): high lutein group
  Interventions: Dietary Supplement: high lutein
- Low lutein zeaxanthin (Experimental): lutein plus zeaxanthin group
  Interventions: Dietary Supplement: lutein plus zeaxanthin
- High zeaxanthin (Experimental): zeaxanthin group
  Interventions: Dietary Supplement: high zeaxanthin
- high lutein zeaxanthin (Experimental): Zeaxanthin plus lutein group
  Interventions: Dietary Supplement: zeaxanthin plus lutein

INTERVENTIONS:
Dietary Supplement: placebo — Placebo, one gelatine capsule containing starch per day, for 96 weeks
  Arms: Placebo
Dietary Supplement: low lutein — one gelatine capsule containing 10mg lutein per day, for 96 weeks
  Arms: Low lutein
Dietary Supplement: high lutein — one gelatine capsule containing 20mg lutein per day, for 96 weeks
  Arms: High lutein
Dietary Supplement: lutein plus zeaxanthin — one gelatine capsule containing 10mg lutein and 10mg zeaxanthin per day, for 96 weeks
  Arms: Low lutein zeaxanthin
Dietary Supplement: high zeaxanthin — one gelatine capsule containing 10mg zeaxanthin per day, for 48 weeks
  Arms: High zeaxanthin
Dietary Supplement: zeaxanthin plus lutein — one gelatine capsule containing 10 mg lutein and 15 mg zeaxanthin per day, for 48 weeks
  Arms: high lutein zeaxanthin

SUMMARY:
This study is to investigate the protective effects of supplemental lutein and zeaxanthin on early age-related macular degeneration (AMD) patients in China.

DETAILED DESCRIPTION:
Early age-related macular degeneration (AMD) is an early hallmark of irreversible vision impairment accompanying with senescence of macular. Given the fact in treatment, prevention strategy is thought to be an efficient and robust approach to diminish early AMD patients in low-income countries, however, feasible cocktail provision in most developing nations remain mysteries. Here we proposed an effective cocktail treatment with different amounts of lutein and zeaxanthin could increase the macular pigment optical density (MPOD) and serum xanthophylls concentrations among randomized Chinese AMD patients; and might improve visual function measured by visual performance indices such as best-spectacle corrected visual acuity (BSCVA), contrast sensitivity (CSF), flash recovery time (FRT), multifocal electroretinogram (mfERG) and microperimetry.

ELIGIBILITY:
Inclusion Criteria:

* aged over 50 years, Chinese of the Han nationality
* diagnosed as age-related macular degeneration
* did not take lutein or zeaxanthin supplements in the past half a year
* good general health
* corrected visual acuity above 0.25 (20/80)
* did not take optical laser or medical treatments

Exclusion Criteria:

* had other ocular diseases, such as glaucoma, macular pucker, optic neuropathy, diabetic retinopathy etc.
* had nervous system diseases, stroke, Type I diabetes
* had diseases effected nutrients absorption, such as Crohn' s disease
* had turbid ocular media or transplanted intraocular lenses
* reported abnormal digestive condition

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Lin, M.M., Principal Investigator — Peking University
Locations (1):
- Haidian District, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ma L, Dou HL, Huang YM, Lu XR, Xu XR, Qian F, Zou ZY, Pang HL, Dong PC, Xiao X, Wang X, Sun TT, Lin XM. Improvement of retinal function in early age-related macular degeneration after lutein and zeaxanthin supplementation: a randomized, double-masked, placebo-controlled trial. Am J Ophthalmol. 2012 Oct;154(4):625-634.e1. doi: 10.1016/j.ajo.2012.04.014. Epub 2012 Jul 25. PMID 22835510

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We added "High Zeaxanthin" and "High Lutein Zeaxanthin" Arms at the seconde year for additional information on the effect of zeaxanthin on MPOD and visual functions. Therefore, we did not measure the changes of serum concentration, and only measured the change of MOPD and visual functions at baseline and 48 weeks, in the two new groups.
Period: Overall Study
Arm/Group | Low Lutein | Placebo | High Lutein | Low Lutein Zeaxanthin | High Zeaxanthin | High Lutein Zeaxanthin
Started | 28 | 28 | 28 | 28 | 28 | 28
Completed | 26 | 28 | 27 | 27 | 28 | 28
Not Completed | 2 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 4 participants was excluded during the analysis since they did not finish the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Lutein | Placebo | High Lutein | Low Lutein Zeaxanthin | High Zeaxanthin | High Lutein Zeaxanthin | Total
Number analyzed (Participants) | 26 | 28 | 27 | 27 | 28 | 28 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (8.3) | 69.0 (7.5) | 69.3 (6.9) | 68.5 (6.9) | 69.7 (5.4) | 69.1 (8.1) | 69.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 13 | 15 | 17 | 15 | 94
  Male | 9 | 11 | 14 | 12 | 11 | 13 | 70
Region of Enrollment [Number; unit: participants]
  China | 26 | 28 | 27 | 27 | 28 | 28 | 164

OUTCOME MEASURES:

1. Primary Outcome: Changes of Macular Pigment Optical Density (MPOD) During 48 Weeks and 2 Years
Description: Macular pigment is found in the center of the retina known as the macula and is made up of the carotenoids lutein and zeaxanthin. This pigment serves to protect the macula from harmful blue light. The MPOD ranges from 0 to 1, with higher scores corresponding with greater density (protection). The autofluorescence picture of subject's macular was analyzed for MPOD values.
  4 participants was excluded during the analysis since they did not finish the intervention. Three did not finish the follow up, while one died from breast cancer.
Time Frame: at baseline and 24 weeks, 48 weeks, 2 years during the intervention
Measure: Mean (Standard Deviation); unit: density units
Arm/Group | Placebo | Low Lutein | High Lutein | Low Lutein Zeaxanthin | High Zeaxanthin | High Lutein Zeaxanthin
Number analyzed (Participants) | 28 | 26 | 27 | 27 | 28 | 28
density units
  baseline | 0.315 (0.144) | 0.307 (0.142) | 0.315 (0.122) | 0.320 (0.118) | 0.327 (0.117) | 0.300 (0.168)
  24 weeks | 0.310 (0.102) | 0.353 (0.125) | 0.395 (0.120) | 0.356 (0.150) | NA (NA) — High zeaxanthin Arm was added after the first 48 weeks to give additional information on the effect of zeaxanthin on MPOD and visual functions, therefore, the change of MPOD from baseline to 48 weeks is all we needed for this purpose. | NA (NA) — "High Lutein Zeaxanthin" Arm was added after the first 48 weeks to give additional information on the effect of zeaxanthin on MPOD and visual functions, therefore, the change of MPOD from baseline to 48 weeks is all we needed for this purpose.
  48 weeks | 0.316 (0.110) | 0.371 (0.188) | 0.424 (0.142) | 0.384 (0.125) | 0.384 (0.139) | 0.383 (0.179)
  2 years | 0.324 (0.163) | 0.442 (0.127) | 0.441 (0.133) | 0.383 (0.149) | NA (NA) — High zeaxanthin Arm was added after the first 48 weeks to give additional information on the effect of zeaxanthin on MPOD and visual functions, therefore, the change of MPOD from baseline to 48 weeks is all we needed for this purpose. | NA (NA) — "High Lutein Zeaxanthin" Arm was added after the first 48 weeks to give additional information on the effect of zeaxanthin on MPOD and visual functions, therefore, the change of MPOD from baseline to 48 weeks is all we needed for this purpose.
Statistical Analysis 1: Comparison: Placebo vs Low Lutein vs High Lutein vs Low Lutein Zeaxanthin; The null hypothesis was no group difference; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Changes of Serum Xanthophylls Concentrations During the Intervention
Description: Changes of serum xanthophylls concentrations measured by high performance liquid chromatograph (HPLC)at baseline and 4, 12, 24 and 48 weeks during the first 48 weeks of intervention.Four participants was excluded during the analysis since they did not finish the intervention. Three did not finish the follow up, while one died from breast cancer.
Time Frame: at baseline and 4, 12, 24 and 48 weeks during the intervention
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Placebo | Low Lutein | High Lutein | Low Lutein Zeaxanthin
Number analyzed (Participants) | 28 | 26 | 27 | 27
μmol/L
  baseline | 0.330 (0.404) | 0.318 (0.251) | 0.301 (0.225) | 0.244 (0.263)
  4 weeks | 0.258 (0.206) | 0.870 (0.573) | 1.041 (0.661) | 0.965 (0.711)
  12 weeks | 0.355 (0.356) | 1.058 (0.571) | 1.450 (0.930) | 1.121 (0.800)
  24 weeks | 0.281 (0.261) | 0.973 (0.618) | 1.450 (0.856) | 1.109 (0.567)
  48 weeks | 0.403 (0.225) | 1.350 (0.503) | 1.876 (0.907) | 1.136 (0.542)
Statistical Analysis 1: Comparison: Placebo vs Low Lutein vs High Lutein vs Low Lutein Zeaxanthin; The null hypothesis was no group difference; Test type: Superiority or Other; p < 0.05, ANOVA

3. Secondary Outcome: Changes of Best-spectacle Corrected Visual Acuity (BSCVA) During the Intervention
Description: best-spectacle corrected visual acuity (BSCVA) measured by ETDRS chart at baseline and 24 weeks, 48 weeks, 2 years during the intervention. Four participants was excluded during the analysis since they did not finish the intervention. Three did not finish the follow up, while one died from breast cancer.
Time Frame: at baseline and 24 weeks, 48 weeks, 2 years during the intervention
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Placebo | Low Lutein | High Lutein | Low Lutein Zeaxanthin | High Zeaxanthin | High Lutein Zeaxanthin
Number analyzed (Participants) | 27 | 26 | 26 | 26 | 27 | 26
letters
  baseline | 53.037 (9.338) | 54.769 (10.285) | 54.539 (8.056) | 56.840 (6.440) | 56.481 (7.073) | 55.038 (7.977)
  24 weeks | 53.444 (12.509) | 54.042 (10.519) | 56.444 (8.617) | 56.160 (14.907) | NA (NA) — High zeaxanthin Arm was added after the first 48 weeks to give additional information on the effect of zeaxanthin on MPOD and visual functions, therefore, the change of BSCVA from baseline to 48 weeks is all we needed for this purpose. | NA (NA) — "High Lutein Zeaxanthin" Arm was added after the first 48 weeks to give additional information on the effect of zeaxanthin on MPOD and visual functions, therefore, the change of BSCVA from baseline to 48 weeks is all we needed for this purpose.
  48 weeks | 53.148 (10.741) | 56.250 (10.920) | 56.846 (10.035) | 60.875 (4.919) | 61.600 (8.093) | 58.500 (9.437)
  2 years | 55.115 (12.385) | 56.840 (7.587) | 56.074 (7.770) | 56.600 (11.839) | NA (NA) — High zeaxanthin Arm was added after the first 48 weeks to give additional information on the effect of zeaxanthin on MPOD and visual functions, therefore, the change of BSCVA from baseline to 48 weeks is all we needed for this purpose. | NA (NA) — "High Lutein Zeaxanthin" Arm was added after the first 48 weeks to give additional information on the effect of zeaxanthin on MPOD and visual functions, therefore, the change of BSCVA from baseline to 48 weeks is all we needed for this purpose.
Statistical Analysis 1: Comparison: Placebo vs Low Lutein vs High Lutein vs Low Lutein Zeaxanthin; The null hypothesis is "no group difference"; Test type: Superiority or Other; p > 0.05, ANOVA

4. Secondary Outcome: Changes of Contrast Sensitivity (CSF) Measured by CSV-100 During the Intervention
Time Frame: at baseline, 24, 48 weeks and 2 years during the intervention
Reporting Status: Not Posted, anticipated posting 2015-12

5. Secondary Outcome: Changes of Flash Recovery Time (FRT) Measured by MDD-2 Macular Adaptometer
Description: Flash recovery time (FRT) was measured by MDD-2 macular adaptometer at baseline, 24, 48 and 96 weeks
Time Frame: at baseline, 24, 48 weeks and 2 years during the intervention
Reporting Status: Not Posted, anticipated posting 2015-12

6. Secondary Outcome: Changes From Baseline in Multifocal Electroretinogram (mfERG) at 48 Weeks
Time Frame: at baseline and 48 weeks during the intervention
Reporting Status: Not Posted, anticipated posting 2015-12

7. Secondary Outcome: Changes From Baseline in Microperimetry (MP) During the Intervention
Description: Microperimetry (MP) was measured by the MP1 Microperimeter
Time Frame: at baseline, 24, 48 weeks and 2 years during the intervention
Reporting Status: Not Posted, anticipated posting 2015-12

8. Secondary Outcome: Changes of Food Pattern From Baseline by Food Frequency Questionnaire During the Intervention
Time Frame: at baseline, 24, 48 weeks and 2 years
Reporting Status: Not Posted, anticipated posting 2015-12

ADVERSE EVENTS:
Time Frame: 2 years, and ask for notable adverse effects for an average interval of 1 month.
Description: 4 participants was excluded during the analysis since they did not finish the intervention. Three did not finish the follow up, while one died from breast cancer. Subjects were encouraged to report any adverse effects immediately, and were asked specifically about adverse events such as carotenoderma every month during visits.
Arm/Group | Placebo | Low Lutein | High Lutein | Low Lutein Zeaxanthin | High Zeaxanthin | High Lutein Zeaxanthin
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26 | 0/27 | 0/27 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/26 | 0/27 | 0/27 | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes